CLINICAL TRIAL: NCT03365063
Title: Integrating Risk-based Care for Patients With Chronic Kidney Disease (CKD) in the Community
Brief Title: Integrating Risk-based Care for Patients With CKD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated early due to COVID-19 restrictions at participating clinics, which made continuation unfeasible.
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Primary Care Sentinel Surveillance Network (Unknown); Canadians Seeking Solutions and Innovations to Overcome Chronic Kidney Disease (Other); Manitoba Primary Care Research Network (MaPCReN) (Unknown); Southern Alberta Primary Care Research Network (SAPCReN) (Unknown)
Responsible Party: Principal Investigator, Navdeep Tangri, Associate Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H2017:050
Record Dates: First submitted 2017-11-28; First posted 2017-12-07 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease
Keywords: Knowledge Translation; Chronic Kidney Disease; Matched Cluster Randomized Trial
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Knowledge Translation Group (Experimental): Primary care clinics receiving the active knowledge translation intervention.
  Interventions: Other: Active Knowledge Translation
- Control Group (No Intervention): Primary care clinics receiving the current standard of care. Information on personalized risk and risk-based referral will not be provided.

INTERVENTIONS:
Other: Active Knowledge Translation — 1. Integration of the KFRE in the CPCSSN DPT - The DPT will report the output from the KFRE for all patients with CKD Stages G3-G5 from the clinic sites. The risk output will include interpretation and automated categorized risk of progression to kidney failure, and will recommend actions based on the KFRE risk based care pathway.
  2. Audit and Feedback - Providers at CPCSSN clinics receive sentinel feedback reports on a panel of chronic conditions and quality improvement targets. The investigators will add CKD to the feedback report for the intervention sites, and provide detailed feedback on the practices' risk profile.
  3. Medical Detailing - The intervention CPCSSN clinics will receive a standardized presentation to clinic staff by the principal investigator, who will provide the evidence for the accuracy of the KFRE and guidance on implementation of a risk based treatment pathway, as well as describe the supporting visual aids.
  Arms: Active Knowledge Translation Group

SUMMARY:
Chronic kidney disease (CKD) and its end stage of kidney failure are major public health problems in Canada and worldwide. In the primary care setting, accurate prediction of the risk of kidney failure in patients with CKD can improve patient provider communication, assist in appropriate nephrology referral, improve dialysis treatment planning, and identify patients who are most likely to benefit from intervention. To aid in accurately predicting the risk of kidney failure requiring dialysis in patients with CKD, the primary investigator has developed and validated the kidney failure risk equation (KFRE), which is increasingly used in nephrology practices across Canada and the United States.

In this current study, a cluster randomized controlled trial (RCT) will be done in collaboration with the Canadian Primary Care Sentinel Surveillance Network (CPCSSN). Primary care clinics that can integrate the KFRE into their electronic medical records will be randomized to receive the intervention (patients and providers receive individualized information explaining kidney failure risk, as well as risk-based criteria for referral, alongside usual care) versus usual care alone (no information on personalized risk and no risk-based referral). In both groups, the investigators will assess management of patients at high risk of kidney failure (patient), timing of referral for patients at high risk of kidney failure (health system), cost of CKD care (health system), CKD-specific health literacy (patient), trust in physician care (patient), and satisfaction with risk prediction tools (provider).

The objective of this research study is to develop, implement, and evaluate tools to guide the care of patients with CKD in the community, including appropriate referral using a risk-based approach. Specifically, this study will address the question: "Does providing patients (and their physicians) with information about their risk of kidney failure improve quality of care, health literacy, and trust in the care they are receiving?"

DETAILED DESCRIPTION:
Patients with CKD and kidney failure have poor outcomes and consume a disproportionate share of health care resources. Therefore, early identification of incident cases by primary care physicians can delay progression and prevent adverse outcomes. However, the correct identification and intervention for patients having reduced kidney function is not necessarily done appropriately in all settings, often resulting in individuals at very low risk of progression being referred to a nephrologist, and in other cases, delayed referral of patients who are at the highest risk of kidney failure.

The investigators propose an integration of the Kidney Failure Risk Equation - a tool that accurately predicts the risk of kidney failure requiring dialysis in patients with CKD - in primary care practices by integrating the tool into existing reporting mechanisms. This will allow the delivery of kidney disease risk information to clinicians as part of a clinical decision aid to guide all aspects of CKD care, including management of vascular risk factors, intensity of follow up, and potential referral for specialist care. Patients and providers will benefit from the ability to share information about CKD, and their individual risk of kidney failure using interactive infographics, thereby improving CKD-specific health literacy.

The investigators will work with the Canadian Primary Care Sentinel Surveillance Network (CPCSSN) to recruit and subsequently randomize 32 clinics to either the intervention or the control group. The clinics randomized to receive the intervention will see patients and providers receiving individualized information explaining kidney failure risk, as well as risk-based criteria for referral, alongside usual care. This will be executed through the integration of the KFRE in the CPCSSN Data Presentation Tool (DPT), audit and feedback, and in-person medical detailing. Clinical decision aids for both patients and physicians to guide CKD care and provide information about prognosis will be provided in the format of a static infographic, video, and interactive website. Those clinics randomized to the control group will receive the current standard of care - information on personalized risk and risk-based referral will not be provided.

Appropriate management of patients at high risk of kidney failure will be determined using information from electronic medical records (EMRs), for all patients with CKD G3-G5 attending each clinic (approximately 13,470 patients from all 32 clinics). Appropriate referral for patients at high risk of kidney failure will be determined through comparison with provincial guidelines. Direct costs of care will be estimated using linkages with provincial administrative data. For those clinics in the intervention group, satisfaction with the risk prediction tools (provider) will be measured using a Likert scale. Additionally,10 patients from each of the 32 clinics will be surveyed about their CKD-specific health literacy and trust in physician care (320 patients in total).

The investigators' hypothesis and specific aims are as follows:

Hypothesis: The investigators hypothesizes that integration of this approach to CKD care can improve the patient-provider dialogue by:

1. Increasing health literacy and trust, and therefore reduce anxiety for those at low risk.
2. Providing early and appropriate referral to nephrology for those at higher risks of kidney failure.

Aim 1 - Determine whether providing patients and primary care providers with a patients' predicted risk for kidney failure and risk-based criteria for referral increases appropriate management of and referral for patients at low and high risk for kidney failure, compared to usual care without personalized risk information.

Aim 2 - Determine whether providing patients with individualized information on their risk of progression increases CKD-specific health literacy and improves trust in the patient-provider relationship.

Aim 3 - Determine the cost-effectiveness of the risk-based care paradigm

Study Design: A matched cluster randomized design of 32 primary care clinics in Manitoba and Alberta, evaluating the feasibility and effectiveness of the integration of the KFRE in the CPCSSN DPT, as well as the efficacy of a KT intervention targeting patients with advanced CKD. The unit of observation will be both at the patient and provider level, and the unit of randomization will be at the level of the clinic.

Team: The investigators' study team includes experts in the clinical epidemiology of CKD and kidney failure, local opinion leaders, as well experts in knowledge translation and cluster randomized design. In addition to the investigators' collaboration with CPCSSN, the investigators are part of and working with the Canadians Seeking Solutions and Innovations to Overcome Chronic Kidney Disease (Can-SOLVE CKD) Network. This network includes individuals with CKD and those affected by CKD (i.e., caregivers, family members, etc.); they are the investigators' patient partners, and will make up the patient engagement panel. They will help guide the study to ensure that its findings are relevant to direct patient care.

Research Significance: Since most patients with CKD are managed in primary care, the next step to reduce the burden of this disease on the population is to implement a strategy for the Kidney Failure Risk Equation to be used in this setting. The investigators believe that the integration of a KFRE based care paradigm can improve management of CKD risk factors and health literacy, and ultimately, downstream patient and health system outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Primary care clinics in Manitoba and Alberta who provide care to adults in the community and use an EMR that can integrate the KFRE and its associated decision aids for CKD management and referral.
* All patients with CKD Stages G3-G5 who attend the 32 clinics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5600 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of CKD patients in each clinic who have albuminuria (albumin-creatinine ratio (ACR)) tested | 1 year after intervention
  This will be determined using data extracted from each clinic's EMR.
The percentage of patients who are appropriately managed with an ACEi or ARB, and who either have CKD and diabetes, or who have CKD and a urine ACR >30 mg/mmol. | 1 year after intervention
  This will be determined using data extracted from each clinic's EMR.

SECONDARY OUTCOMES:
Diabetes management for CKD patients | 1 year after intervention
  Measured as the proportion of CKD patients who have a hemoglobin A1C in target (i.e. <8.5%), as well as the proportion of individuals who have been prescribed an SGLT2 inhibitor.
Hypertension management for CKD patients | 1 year after intervention
  Measured as the proportion of CKD patients who have a normal blood pressure (BP), taken as part of regular clinic visit (office BP <130/80 for patients with diabetes, 140/90 for those without).
Management of cardiovascular risk factors for CKD patients | 1 year after intervention
  Measured as the proportion of CKD patients who have a statin prescription listed on their EMR.
Appropriate medication usage | 1 year after intervention
  Measured as the proportion of CKD patients who have been prescribed a non-steroidal anti-inflammatory drug (NSAID).
eGFR function for CKD patients | 2 years after intervention
  Measured as the proportion of CKD patients who have a >30% decline in eGFR function.
Appropriate referral for patients at high risk for kidney failure | 1 year after intervention
  Determined through comparisons with provincial guidelines.
Total Health Care Costs | 1 year after intervention
  Direct health care costs will be estimated for both groups of patients taking a health care payor perspective, and estimated using linkages with provincial administrative data.
Clinical provider's satisfaction with the risk prediction tools and clinical decision aids. | 6 months after intervention
  Measured by the number of points as a result of the clinical providers' answers on a Likert scale.
Patient's CKD-specific health literacy | 6 months after intervention
  Measured by the number of points as a result of participants' answers to the validated Kidney Knowledge Survey (KiKS).
Patient's trust in physician care | 6 months after intervention
  Measured by the number of points as a result of participants' answers to the validated Trust in Physician Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Navdeep Tangri, MD PhD FRCPC, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - Southern Alberta Primary Care Research Network (SAPCReN), Calgary, Alberta
  - University of Manitoba, Winnipeg, Manitoba

REFERENCES:
- [Background] Harasemiw O, Drummond N, Singer A, Bello A, Komenda P, Rigatto C, Lerner J, Sparkes D, Ferguson TW, Tangri N. Integrating Risk-Based Care for Patients With Chronic Kidney Disease in the Community: Study Protocol for a Cluster Randomized Trial. Can J Kidney Health Dis. 2019 May 29;6:2054358119841611. doi: 10.1177/2054358119841611. eCollection 2019. PMID 31191908
- [Background] Bello AK, Ronksley PE, Tangri N, Kurzawa J, Osman MA, Singer A, Grill A, Nitsch D, Queenan JA, Wick J, Lindeman C, Soos B, Tuot DS, Shojai S, Brimble S, Mangin D, Drummond N. Prevalence and Demographics of CKD in Canadian Primary Care Practices: A Cross-sectional Study. Kidney Int Rep. 2019 Jan 21;4(4):561-570. doi: 10.1016/j.ekir.2019.01.005. eCollection 2019 Apr. PMID 30993231
- [Background] Bello AK, Ronksley PE, Tangri N, Kurzawa J, Osman MA, Singer A, Grill AK, Nitsch D, Queenan JA, Wick J, Lindeman C, Soos B, Tuot DS, Shojai S, Brimble KS, Mangin D, Drummond N. Quality of Chronic Kidney Disease Management in Canadian Primary Care. JAMA Netw Open. 2019 Sep 4;2(9):e1910704. doi: 10.1001/jamanetworkopen.2019.10704. PMID 31483474
- See also: Study Website — http://www.kidneyfailurerisk.com